CLINICAL TRIAL: NCT03118934
Title: Assessing Fitting Guides in Alcon Multifocal Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CLK027-P001
Record Dates: First submitted 2017-04-11; First posted 2017-04-18 (Actual); Results first posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Presbyopia; Refractive Errors
Keywords: contact lenses; presbyopia; multifocal
MeSH Terms: conditions — Presbyopia; Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects are unmasked to the study lenses that are dispensed, but will be masked to the fitting guides used to fit each eye.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- AOA MF (Experimental): Lotrafilcon B multifocal contact lenses worn bilaterally (in both eyes) for 10 ± 3 days
  Interventions: Device: Lotrafilcon B multifocal contact lenses
- DACP MF (Experimental): Nelfilcon A multifocal contact lenses worn bilaterally for 10 ± 3 days
  Interventions: Device: Nelfilcon A multifocal contact lenses
- DT1 MF (Experimental): Delefilcon A multifocal contact lenses worn bilaterally for 10 ± 3 days
  Interventions: Device: Delefilcon A multifocal contact lenses

INTERVENTIONS:
Device: Lotrafilcon B multifocal contact lenses — Contact lenses for near, intermediate, and distance correction worn on a daily wear basis and cared for with participant's habitual lens care solution
  Other Names: AIR OPTIX AQUA® Multifocal
  Arms: AOA MF
Device: Nelfilcon A multifocal contact lenses — Contact lenses for near, intermediate, and distance correction worn on a daily disposable basis (removed every night and discarded) with a new pair of study lenses every morning
  Other Names: DAILIES® AquaComfort Plus® Multifocal
  Arms: DACP MF
Device: Delefilcon A multifocal contact lenses — Contact lenses for near, intermediate, and distance correction worn on a daily disposable basis (removed every night and discarded) with a new pair of study lenses every morning
  Other Names: DAILIES TOTAL1® Multifocal
  Arms: DT1 MF

SUMMARY:
The purpose of this study is to compare an alternative fitting guide to a current fitting guide for optimizing contact lens parameters and determining contact lens prescription.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent;
* Normal eyes;
* Current full-time soft contact lens wearer needing presbyopia correction;
* Willing to wear lenses for a minimum of five days per week, six hours per day, and attend all study visits;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Use of systemic or ocular medications for which contact lens wear could be contraindicated as determined by the Investigator;
* Eye conditions (past or present) as specified in the protocol;
* Currently wearing Alcon multifocal (MF) contact lenses;
* Only one eye with functional vision;
* Contact lens wear in one eye only;
* Use of mechanical eyelid therapy or eyelid scrubs within 14 days before Visit 1 and not willing to discontinue during the study;
* Other protocol-defined exclusion criteria may apply.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Manager, Vision Care, Study Director — Alcon Research
Locations (19):
- United States (13):
  - Alcon Investigative Site, Phoenix, Arizona
  - Alcon Investigative Site, San Diego, California
  - Alcon Investigative Site, Pensacola, Florida
  - Alcon Investigative Site, Tallahassee, Florida
  - Alcon Investigative Site, Pittsburg, Kansas
  - Alcon Investigative Site, Shawnee Mission, Kansas
  - Alcon Investigative Site, Ann Arbor, Michigan
  - Alcon Investigative Site, Eden Prairie, Minnesota
  - Alcon Investigative Site, Medina, Minnesota
  - Alcon Investigative Site, Raytown, Missouri
  - Alcon Investigative Site, Powell, Ohio
  - Alcon Investigative Site, Warwick, Rhode Island
  - Alcon Investigative Site, Memphis, Tennessee
- Canada (3):
  - Alcon Investigative Site, Burnaby, British Columbia
  - Alcon Investigative Site, Toronto, Ontario
  - Alcon Investigative Site, Toronto
- United Kingdom (3):
  - Alcon Investigative Site, Coventry
  - Alcon Investigative Site, Hereford
  - Alcon Investigative Site, Monmouth

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 20 investigational sites located in the United States (14), United Kingdom (3), and Canada (3).
Pre-assignment Details: Of the 188 enrolled subjects, 6 were exited prior to trial fit. This reporting group includes all subjects randomized and trial fit, as randomized (182). Safety Analysis Set is reported as exposed.
Groups:
- AOA MF - Alternative: Bilaterally (in both eyes) fitted using alternative fitting guide; lotrafilcon B multifocal contact lenses worn bilaterally for 10 ± 3 days
- DACP MF - Alternative: Bilaterally fitted using alternative fitting guide; nelfilcon A multifocal contact lenses worn bilaterally for 10 ± 3 days
- DT1 MF - Alternative: Bilaterally fitted using alternative fitting guide; delefilcon A multifocal contact lenses worn bilaterally for 10 ± 3 days
- AOA MF - Current: Bilaterally fitted using current fitting guide; lotrafilcon B multifocal contact lenses worn bilaterally (in both eyes) for 10 ± 3 days
- DACP MF - Current: Bilaterally fitted using current fitting guide; nelfilcon A multifocal contact lenses worn bilaterally for 10 ± 3 days
- DT1 MF - Current: Bilaterally fitted using current fitting guide; delefilcon A multifocal contact lenses worn bilaterally for 10 ± 3 days
Period: Overall Study
Arm/Group | AOA MF - Alternative | DACP MF - Alternative | DT1 MF - Alternative | AOA MF - Current | DACP MF - Current | DT1 MF - Current
Started (Randomized and trial fit, as randomized) | 34 | 31 | 34 | 29 | 29 | 25
Safety Analysis Set (All subjects/eyes exposed to study lenses, except those used for trial fit at Visit 1, as exposed) | 34 | 29 | 34 | 29 | 26 | 25
Completed (Completed, as randomized) | 34 | 30 | 33 | 28 | 27 | 23
Not Completed | 0 | 1 | 1 | 1 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Discontinued prior to exposure | 0 | 1 | 1 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set. Baseline data analyzed based on study lens.
Groups:
- AOA MF: Lotrafilcon B multifocal contact lenses worn bilaterally for 10 ± 3 days
- Total: Total of all reporting groups
Arm/Group | AOA MF | DACP MF | DT1 MF | Total
Number analyzed (Participants) | 63 | 55 | 59 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (6.9) | 50.1 (6.7) | 50.1 (6.7) | 50.3 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 46 | 52 | 149
  Male | 12 | 9 | 7 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 55 | 48 | 51 | 154
  Black or African American | 2 | 4 | 0 | 6
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 2 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Other | 1 | 1 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Trial Lenses Needed to Fit Each Eye
Description: The Investigator used a multi-focal contact lens fitting guide to determine which study lens to fit
Time Frame: VIsit 1/Day 1
Population: This analysis population includes all subjects randomized or assigned to study lenses as applicable, and exposed to study lenses including trial fit at Visit 1 (Full Analysis Set).
Measure: Mean (Standard Deviation); unit: lenses
Units Other Than Participants: Eyes
Groups:
- Alternative: Bilaterally fitted with trial lenses using the alternative fitting guide
- Current: Bilaterally fitted with trial lenses using the current fitting guide
Arm/Group | Alternative | Current
Number analyzed (Participants) | 99 | 83
Number analyzed (Eyes) | 198 | 166
lenses | 1.2 (0.5) | 1.4 (0.5)
Statistical Analysis 1: Comparison: Alternative vs Current; Test type: Non-Inferiority — The pre-specified non-inferiority margin is 0.5. With a sample size of 80/group, there was approximately 83% power to reject the null hypothesis of inferiority in fit with assumed standard deviation of 0.6 and expected difference of 0.25 (one-sided alpha=0.05); LSM Difference = -0.2, 95% CI 1-sided [upper limit -0.1], Standard Error of Mean 0.06

ADVERSE EVENTS:
Time Frame: Screening/Fitting through study completion, a maximum of 33 days.
Description: Adverse Events (AE) were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. Safety Analysis Set, as exposed, which is different than "as randomized" due to subjects not following the assigned randomization. "At risk" population for ocular AEs is reported in units of eyes.
Groups:
- AOA MF Ocular: Eyes exposed to AIR OPTIX AQUA® Multifocal (AOA MF) contact lenses
- AOA MF Nonocular: Subjects exposed to AOA MF contact lenses
- DACP MF Ocular: Eyes exposed to DAILIES® AquaComfort Plus® Multifocal (DACP MF) contact lenses
- DACP MF Nonocular: Subjects exposed to DACP MF contact lenses
- DT1 MF Ocular: Eyes exposed to DAILIES TOTAL1® Multifocal (DT1 MF) contact lenses
- DT1 MF Nonocular: Subjects exposed to DT1 MF contact lenses
Arm/Group | AOA MF Ocular | AOA MF Nonocular | DACP MF Ocular | DACP MF Nonocular | DT1 MF Ocular | DT1 MF Nonocular
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/63 | 0/110 | 0/55 | 0/118 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/63 | 0/110 | 0/55 | 0/118 | 0/59
Other Adverse Events (participants affected / at risk) | 0/126 | 0/63 | 0/110 | 0/55 | 0/118 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/34/NCT03118934/SAP_000.pdf
  • Study Protocol (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/34/NCT03118934/Prot_001.pdf